CLINICAL TRIAL: NCT06215729
Title: The Therapeutic Effect of Computer-assisted Cognitive Function Training on Cognitive Dysphagia After Stroke: A Randomized Controlled Study
Brief Title: The Therapeutic Effect of Computer-assisted Cognitive Function Training on Cognitive Dysphagia After Stroke
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: ethical issues
Sponsor: Zeng Changhao (Other)
Responsible Party: Sponsor-Investigator, Zeng Changhao, Research Director, People's Hospital of Zhengzhou University
Organization: People's Hospital of Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-KY-1229
Record Dates: First submitted 2024-01-11; First posted 2024-01-22 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Dysphagia; Cognitive Impairment; Stroke
MeSH Terms: conditions — Deglutition Disorders; Cognitive Dysfunction; Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the experimental group (Experimental): In this study, each patient received a continuous 15-day treatment. During the treatment, both groups of patients received routine rehabilitation treatment. The experimental group additionally underwent computer-assisted cognitive training, which generated training content of corresponding difficulty based on the patient's cognitive impairment assessment results. The training was conducted seven days a week, once a day, for a duration of 30-45 minutes per session.
  Interventions: Behavioral: routine rehabilitation treatment; Behavioral: Computer-assisted Cognitive Function Training
- the control group (Active Comparator): In this study, each patient received a continuous 15-day treatment. During the treatment, both groups of patients received routine rehabilitation treatment.The control group was given conventional cognitive training.
  Interventions: Behavioral: routine rehabilitation treatment; Behavioral: conventional cognitive training

INTERVENTIONS:
Behavioral: routine rehabilitation treatment — The routine rehabilitation treatment included intervention for risk factors (such as blood pressure, blood lipids, and blood glucose control, restriction of smoking and alcohol, exercise, etc.) Besides, the patients with stable vital signs were scheduled for specialized rehabilitation training upon enrollment, and targeted rehabilitation programs were selected, conducted by experienced rehabilitation therapists.
Behavioral: conventional cognitive training — including Memory training, attention training, and executive function training were conducted 2-5 times per week, lasting for 30-60 minutes each session, based on the patient's condition.
  Arms: the control group
Behavioral: Computer-assisted Cognitive Function Training — Based on the patient's cognitive impairment assessment results, the training content includes Attention game training, Executive function program training, Logical reasoning training, Agility training, Memory training. The training is conducted seven days a week, once a day, for a duration of 30-45 minutes per session
  Arms: the experimental group

SUMMARY:
This is a multicenter randomized controlled study. The study recruited stroke patients with mild cognitive impairment and dysphagia who were undergoing inpatient rehabilitation treatment in three hospitals in mainland China as the participants (study subjects). The study duration for each participant was 15 days. The subjects were randomly divided into an experimental group and a control group. During the treatment, all patients received routine rehabilitation treatment. In addition, patients in the control group received conventional cognitive training, while patients in the experimental group received computer-assisted cognitive training.

DETAILED DESCRIPTION:
Computer-assisted cognitive training is a rehabilitation method that uses computer technology and psychological principles to promote the recovery of cognitive function.This is a multicenter randomized controlled study. The study recruited stroke patients with mild cognitive impairment and dysphagia who were undergoing inpatient rehabilitation treatment in three hospitals in mainland China as the participants (study subjects). The study duration for each participant was 15 days. The subjects were randomly divided into an experimental group and a control group. During the treatment, all patients received routine rehabilitation treatment. In addition, patients in the control group received conventional cognitive training, while patients in the experimental group received computer-assisted cognitive training.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Meeting the diagnostic criteria for traumatic brain injury, confirmed by magnetic resonance imaging or CT scan.
* Montreal Cognitive Assessment score < 26 and > 18 (adjusted by 1 point if the educational level is high school graduation or above).
* Confirmed swallowing disorder through Fiberoptic Endoscopic Examination of Swallowing.
* Duration of illness greater than three months.
* Patients or their family members are aware of and consent to participate in the study.

Exclusion Criteria:

* Presence of other intracranial lesions, such as stroke.
* Cognitive impairment caused by other diseases.
* Mental abnormalities.
* Inability to complete treatment and assessments due to other impairments.
* Concurrent severe injuries.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-04-15 (Estimated); Study Completion 2024-04-15 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment | day 1 and day 15
  The Montreal Cognitive Assessment is used for assessing cognitive function.The total score on the test is 30, the higher scores indicating the higher cognitive function

SECONDARY OUTCOMES:
The coordination of swallowing | day 1 and day 15
  Observation of the coordination of laryngeal and vocal fold movements. Results are categorized as normal/abnormal.
Penetration-Aspiration Scale | day 1 and day 15
  Penetration-Aspiration Scale was used to assess dysphagia under Videofluoroscopic Swallowing Study, primarily evaluating the extent to which fluid food entered the airway and caused penetration or aspiration during the swallowing process. As the level increased, the severity of dysphagia also increased.
Swallowing duration | day 1 and day 15
  The time duration that the patient swallowed the contrast agent under Videofluoroscopic Swallowing Study the was recorded.Unit: seconds.
Swallowing reflex | day 1 and day 15
  Observation of the ability to initiate swallowing movements during eating, manifested by the white-out phenomenon seen under flexible laryngoscopy. Results are categorized as normal or abnormal.

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Master, Principal Investigator — Site Coordinator of United Medical Group located in Miami
Locations (1):
- Zheng da yi fu yuan hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No